CLINICAL TRIAL: NCT04378127
Title: Educational Therapy in Parkinson's Disease (PD): A Non-pharmacological Interventional, Multicentric, Randomized Controlled Trial.
Brief Title: Mister Parkinson: Educational Therapy in Parkinson's Disease (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MisterParkinson
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; burden; caregiver; educational program
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This was a single-blind,multicentric, prospective, randomized study comparing two arms: an intervention group undergoing a structured educational program associated to standard care and a control group who solely continued with traditional medical care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- educational program + traditional medical care (Experimental): The educational program consisted of six thematic meetings of 3 hours each, which a 15-minute interval every hour. Each meeting had a key topic and was divided in a teaching session and in a practical session with individual training of both, subject and caregiver. Every lecture was held by a movement disorders specialist with particular expertise in each field of discussion and the content of each lessons (slides, flyers, questionnaires) was adapted to fit the audience.
  Interventions: Other: Educational program
- traditional medical care (No Intervention): traditional medical care

INTERVENTIONS:
Other: Educational program — The educational program consisted of six thematic meetings of 3 hours each, which a 15-minute interval every hour. Each meeting had a key topic and was divided in a teaching session and in a practical session with individual training of both, subject and caregiver. Every lecture was held by a movement disorders specialist with particular expertise in each field of discussion and the content of each lessons (slides, flyers, questionnaires) was adapted to fit the audience.
  Arms: educational program + traditional medical care

SUMMARY:
Parkinson's disease is multidimensional disorders characterized by motor and non-motor symptoms such as behavioral and psychological symptoms, autonomic disturbances and other non-motor symptoms. These can contribute to the burden of the disease on patients and their caregivers, and often remain unrecognized and untreated.

This was a single-blind,multicentric, prospective, randomized study comparing two arms: an intervention group undergoing a structured educational program associated to standard care and a control group who solely continued with traditional medical care.

DETAILED DESCRIPTION:
Parkinson's disease is multidimensional disorders characterized by motor and non-motor symptoms such as behavioral and psychological symptoms, autonomic disturbances and other non-motor symptoms. A multidisciplinary and comprehensive approach, based on the chronic care model, is considered the best way to manage motor and non-motor symptoms of the disease, although this model of care is still not standardized and previous trials showed conflicting results.

The study planned to enrol 40 advanced PD patients and related caregivers for each investigational site. This was a single-blind,multicentric, prospective, randomized study comparing two arms: an intervention group undergoing a structured educational program associated to standard care and a control group who solely continued with traditional medical care.

The educational program consisted of six thematic meetings of 3 hours each, which a 15-minute interval every hour. Each meeting had a key topic and was divided in a teaching session and in a practical session with individual training of both, subject and caregiver. Every lecture was held by a movement disorders specialist with particular expertise in each field of discussion and the content of each lessons (slides, flyers, questionnaires) was adapted to fit the audience.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease (according to UK Brain Bank criteria)
* being aged 20-80 years
* being able to complete questionnaires
* having no severe cognitive impairment (mini-mental state examination ≥24)
* having a stable caregiver

Exclusion Criteria:

* atypical parkinsonian
* severe comorbidity significantly interfering with quality of life

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
OFF hours | through study completion, an average of 1 year
  The primary outcome was change from baseline to end of study in the mean daily OFF hours evaluated with the Hauser diary.
  Expected increase in the mean time spent in ON in at least 50% of treated patients (OR ≥1.5) compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: fabrizio stocchi, md phd, Principal Investigator — IRCCS San Raffaele

IPD SHARING:
Plan to Share IPD: Yes
after the end of sudy
Supporting Information: Study Protocol
Time Frame: after the end of study
Access Criteria: request by email

REFERENCES:
- [Derived] De Pandis MF, Torti M, Rotondo R, Iodice L, Levi Della Vida M, Casali M, Vacca L, Viselli F, Servodidio V, Proietti S, Stocchi F. Therapeutic education for empowerment and engagement in patients with Parkinson's disease: A non-pharmacological, interventional, multicentric, randomized controlled trial. Front Neurol. 2023 Apr 18;14:1167685. doi: 10.3389/fneur.2023.1167685. eCollection 2023. PMID 37144003